CLINICAL TRIAL: NCT02561715
Title: Lack of Awareness of Symptoms (Anosognosia) in PD: An Observational Study to Examine the Effects of Anosognosia on Self-Reported Quality of Life for People With Parkinson's
Brief Title: Lack of Awareness of Symptoms (Anosognosia) in PD: An Observational Study for People With Parkinson's
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RG_14-096
Record Dates: First submitted 2015-08-28; First posted 2015-09-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's; Anosognosia
Keywords: Parkinson's; Anosognosia; DBS; Deep Brain Surgery
MeSH Terms: conditions — Parkinson Disease; Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Questionnaires — Pre and post deep brain surgery questionnaires

SUMMARY:
Anosognosia is a recognised condition for people with Parkinson's, and is the result of physiological damage on brain structure.

Surgical Parkinson Disease Nurse Specialists have noticed that when reviewing the pre-surgery videos 12 months post-DBS, patients have forgotten and are shocked at how bad their symptoms were prior to surgery (personal communication), which may not be reflected in the change in QoL reported.

This lack of awareness, while possibly helpful in everyday life, may lead to effective treatments looking ineffective, or the benefits in QoL of effective treatment appearing reduced. This confound may not only reduce the apparent effectiveness but also the related cost-effectiveness of treatment. As cost-effectiveness is determined by both size and longevity of an effect, current methods of capturing these data may be suboptimal.

DETAILED DESCRIPTION:
The overarching aim of this project is to identify coping mechanisms and pathological lack of self-awareness and the impact they are likely to have on patient reported quality of life (QoL) outcome measures for a chronic condition.

This will be an observational study, a case series of approx. 10 to 20 patients. These patients will be recruited over a 6 month period from the Queen Elizabeth Hospital, Birmingham and will be informed of the study during their routine pre-surgical visit.

Patients will be eligible if they are about to undergo DBS at Queen Elizabeth Hospital. If the participant has a carer, who is also willing to participate, they may also join the study. Patients will be excluded if they are unable to complete questionnaires in English.

Once recruited and following consent, a patient will complete a brief battery of questionnaires both self-reported and clinician rated prior to surgery and at their 6 month post op visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's as defined by the UK PDS Brain Bank Criteria

Exclusion Criteria:

* Unable to complete questionnaires in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's due for deep brain surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Improvement of ability to recall extent of condition | 9 months
  Person with Parkinson's specific quality of life using the Parkinson's Disease Questionnaire for both participant and carer.

SECONDARY OUTCOMES:
Clinician's Rating Scale for Evaluating Impaired Self Awareness and Denial of Disability after Brain Injury adapted for use with PD patients.after Brain Injury, adapted for use with Parkinson's Disease patients | 9 months
  Participants self-awareness of their Parkinson's
Patient Generated Index | 9 months
  Quality of life measure
Abnormal Involuntary Movement Scale | 9 months
  Occurrence of tardive dyskinesia
Patient Competency Rating Scale | 9 months
  Evaluation of self-awareness following traumatic brain injury
Grooved peg board test | 9 months
  Measuring motor performance
The tapping test | 9 months
  Measuring motor control
Unified Parkinson's Disease Rating Scale | 9 months
  Rating the extent of the participant's Parkinson's
Mini Mental State Exam | 9 months
  Measure of cognitive impairment
Parkinson's' Disease Questionnaire | 9 months
  PDQ-39 (Carer)

CONTACTS AND LOCATIONS:
Overall Officials: Hardev Pall, MD, Principal Investigator — Queen Elizabeth Medical Centre, Birmingham, UK
Locations (1):
- Queen Elizabeth Hospital, Birmingham, United Kingdom